CLINICAL TRIAL: NCT05958433
Title: Preoperative Rehabilitation With Stoma Appliance in Colorectal Cancer Patients, A Randomized Controlled Trial
Brief Title: Preoperative Rehabilitation With Stoma Appliance in Colorectal Cancer Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mariana kamal, principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: PRWSACRC
Record Dates: First submitted 2023-07-05; First posted 2023-07-24 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Rehabilitation
MeSH Terms: interventions — Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- standard postoperative education. (Active Comparator): These patients will receive stoma care and stoma education beginning on postoperative day1.
  Interventions: Behavioral: Rehabilitation with stoma appliance
- preoperative rehabilitation group (Experimental): The rehabilitation group will receive preoperative stoma education in addition
  Interventions: Behavioral: Rehabilitation with stoma appliance

INTERVENTIONS:
Behavioral: Rehabilitation with stoma appliance — The rehabilitation group will receive preoperative stoma education in addition, a water-filled ostomy appliance (50-100 ml) will be attached 48 hours before surgery. These pouches will not be removed until surgery, and the EST nurse will teach the patients preoperatively how to manage the ostomy appliance with similar standards as described in the usual postoperative stoma care.

SUMMARY:
This is a randomized, controlled trial aiming to assess the effects of preoperative education using stoma appliance on stoma self-care, quality of life, anxiety, and depression levels in colorectal cancer patients with a stoma.

DETAILED DESCRIPTION:
Colorectal cancer is third cancer worldwide after breast and lung cancer accounting for 10% of all cancer cases and 9.4% of cancer deaths. Over 2.2 million new colorectal cancer cases and 1.8 million deaths have been estimated to occur in 2020. In Egypt, it is the seventh cancer, accounting for 3.9% of all cancers, with about 5,000 new cases annually.

Colorectal resections are often associated with temporary or permanent stoma formations. In the United Kingdom it is estimated that more than 20,000 new stomas are created each year, 11,800 of them were colostomies. About one-half of the stoma was permanent. The formation of a stoma is associated with psychologic morbidity, which can be reduced with preoperative and postoperative patient education and psychologic support.

Living with a stoma is a challenging situation for various reasons including uncontrolled gas passage through it, diarrhea, odor, and leakage around the stoma or appliance. It would take several months for the patients to adjust to this difficult time. At that point, the patient's Quality of life becomes essential for the remaining time.

Ostomy formation is one of the therapeutic procedures performed to manage bowel dysfunction due to various reasons; however, it affects quality of life of patients. World health organization defines QOL as an individual's perspective of his/her health status concerning a few aspects- physical, psychological, economic, social, and environmental.

A stoma influences the physical, mental, emotional, and social life of the patient significantly. A good quality of life is essential to achieve a comprehensive approach to treating patients. A study done in China to assess stoma related quality of life using a stoma self-care agency scale and health hope index showed that patients had difficulties in work and social institutions. Additional concerns pointed out were sexuality, body image and the stoma itself. A long-term effect on the quality of life of members of the United Ostomy Association of America after 5 years of ostomy surgery was assessed using a questionnaire. Their report has shown that patients feel better as they live longer with the stoma. Research done on Iranian by ostomy society has shown that factors such as the type of ostomy, the underlying disease that had led to the stoma formation, depression after ostomy, dissatisfaction with sexual activities, a problem with the location of ostomy and change in clothing style affected the Quality of Life.

Ostomies can lead to intensified distress and suffering in patients because of skin irritation (76%), pouch leakage (62%), offensive odor (59%), reduction in pleasurable activities (54%), and depression/anxiety (53%). In such circumstances, it is worthwhile to assess the quality of life in the evaluation of the outcomes of various therapeutic procedures along with their final impact on patients' lives. Quality of care and training provided to patients can be associated with their subsequent quality of life. The main aim of this study is to assess the effects of preoperative education on stoma self-care, quality of life, Anxiety, and depression levels in colorectal cancer patients with a stoma.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective operable colorectal resections that would require the formation of a temporary or permanent stoma.
* Patients who were likely to be self-sufficient in managing their stoma pouching system after surgery.

Exclusion Criteria:

1. Those who undergo emergency surgery
2. Disoriented patients who cannot cooperate.
3. Patients with psychiatric disease.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2023-08 (Estimated); Primary Completion 2024-08 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
duration of hospital stay | 1 year
  Compare duration from surgery until independent stoma self-care between preoperative rehabilitation using a stoma appliance group and traditional care group.

SECONDARY OUTCOMES:
Assess anxiety and depression | 9 monthes
  Assess anxiety and depression according to HADS (Hospital Anxiety and Depression Scale).
  0-7 normal 8-10 border line abnormal 11-21 abnormal
assess the effects of preoperative education using stoma appliance on quality of life in colorectal cancer patients with a stoma | 11 months
  Assess the quality of life of those patients including physical, social/family, emotional, functional wellbeing, using FACT-C version 4 (Functional Assessment of Cancer Therapy-Colorectal) questionnaire.
  recall period past 7 days response scale 5point Likert-type scale total a FACT-C score (functional assessment of cancer therapy -colorectal) range 0-136 the higher the score the better the quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Nelly AliEldien, proffesor, Study Chair — Prof. Biostatistics & Cancer Epidemiology National Cancer Institute, Cairo University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Background] Archambault AN, Su YR, Jeon J, Thomas M, Lin Y, Conti DV, Win AK, Sakoda LC, Lansdorp-Vogelaar I, Peterse EFP, Zauber AG, Duggan D, Holowatyj AN, Huyghe JR, Brenner H, Cotterchio M, Bezieau S, Schmit SL, Edlund CK, Southey MC, MacInnis RJ, Campbell PT, Chang-Claude J, Slattery ML, Chan AT, Joshi AD, Song M, Cao Y, Woods MO, White E, Weinstein SJ, Ulrich CM, Hoffmeister M, Bien SA, Harrison TA, Hampe J, Li CI, Schafmayer C, Offit K, Pharoah PD, Moreno V, Lindblom A, Wolk A, Wu AH, Li L, Gunter MJ, Gsur A, Keku TO, Pearlman R, Bishop DT, Castellvi-Bel S, Moreira L, Vodicka P, Kampman E, Giles GG, Albanes D, Baron JA, Berndt SI, Brezina S, Buch S, Buchanan DD, Trichopoulou A, Severi G, Chirlaque MD, Sanchez MJ, Palli D, Kuhn T, Murphy N, Cross AJ, Burnett-Hartman AN, Chanock SJ, de la Chapelle A, Easton DF, Elliott F, English DR, Feskens EJM, FitzGerald LM, Goodman PJ, Hopper JL, Hudson TJ, Hunter DJ, Jacobs EJ, Joshu CE, Kury S, Markowitz SD, Milne RL, Platz EA, Rennert G, Rennert HS, Schumacher FR, Sandler RS, Seminara D, Tangen CM, Thibodeau SN, Toland AE, van Duijnhoven FJB, Visvanathan K, Vodickova L, Potter JD, Mannisto S, Weigl K, Figueiredo J, Martin V, Larsson SC, Parfrey PS, Huang WY, Lenz HJ, Castelao JE, Gago-Dominguez M, Munoz-Garzon V, Mancao C, Haiman CA, Wilkens LR, Siegel E, Barry E, Younghusband B, Van Guelpen B, Harlid S, Zeleniuch-Jacquotte A, Liang PS, Du M, Casey G, Lindor NM, Le Marchand L, Gallinger SJ, Jenkins MA, Newcomb PA, Gruber SB, Schoen RE, Hampel H, Corley DA, Hsu L, Peters U, Hayes RB. Cumulative Burden of Colorectal Cancer-Associated Genetic Variants Is More Strongly Associated With Early-Onset vs Late-Onset Cancer. Gastroenterology. 2020 Apr;158(5):1274-1286.e12. doi: 10.1053/j.gastro.2019.12.012. Epub 2019 Dec 19. PMID 31866242
- [Background] Chaudhri S, Brown L, Hassan I, Horgan AF. Preoperative intensive, community-based vs. traditional stoma education: a randomized, controlled trial. Dis Colon Rectum. 2005 Mar;48(3):504-9. doi: 10.1007/s10350-004-0897-0. PMID 15768181
- [Background] Zewude WC, Derese T, Suga Y, Teklewold B. Quality of Life in Patients Living with Stoma. Ethiop J Health Sci. 2021 Sep;31(5):993-1000. doi: 10.4314/ejhs.v31i5.11. PMID 35221616
- [Background] Anaraki F, Vafaie M, Behboo R, Maghsoodi N, Esmaeilpour S, Safaee A. Quality of life outcomes in patients living with stoma. Indian J Palliat Care. 2012 Sep;18(3):176-80. doi: 10.4103/0973-1075.105687. PMID 23439841
- [Background] Richbourg L, Thorpe JM, Rapp CG. Difficulties experienced by the ostomate after hospital discharge. J Wound Ostomy Continence Nurs. 2007 Jan-Feb;34(1):70-9. doi: 10.1097/00152192-200701000-00011. PMID 17228210
- [Background] Krouse RS, Grant M, Rawl SM, Mohler MJ, Baldwin CM, Coons SJ, McCorkle R, Schmidt CM, Ko CY. Coping and acceptance: the greatest challenge for veterans with intestinal stomas. J Psychosom Res. 2009 Mar;66(3):227-33. doi: 10.1016/j.jpsychores.2008.09.009. Epub 2009 Jan 16. PMID 19232235
- [Background] Prieto L, Thorsen H, Juul K. Development and validation of a quality of life questionnaire for patients with colostomy or ileostomy. Health Qual Life Outcomes. 2005 Oct 12;3:62. doi: 10.1186/1477-7525-3-62. PMID 16219109
- [Background] Bocerean C, Dupret E. A validation study of the Hospital Anxiety and Depression Scale (HADS) in a large sample of French employees. BMC Psychiatry. 2014 Dec 16;14:354. doi: 10.1186/s12888-014-0354-0. PMID 25511175